CLINICAL TRIAL: NCT00294658
Title: A Multi-Center, Single-Blind, Randomized Study Comparing Thymectomy to No Thymectomy in Non-Thymomatous Myasthenia Gravis (MG) Patients Receiving Prednisone
Brief Title: Thymectomy Trial in Non-Thymomatous Myasthenia Gravis Patients Receiving Prednisone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gary Cutter, PhD, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NS050733; 1U01NS042685-01A2 (NIH); CRC (Other: NINDS)
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; thymectomy; prednisone; corticosteroid; extended transsternal thymectomy; ETTX; MG; thymus; thymoma
MeSH Terms: conditions — Myasthenia Gravis; Thymoma | interventions — Thymectomy; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymectomy plus prednisone (Active Comparator): Procedure: Extended Transsternal Thymectomy plus prednisone treatment
  Interventions: Procedure: thymectomy plus prednisone
- Prednisone alone (Placebo Comparator): Drug: prednisone alone protocol
  Interventions: Drug: prednisone alone

INTERVENTIONS:
Procedure: thymectomy plus prednisone — The thymectomy will be performed as soon as possible after randomization.
  Other Names: Extended transsternal thymectomy plus prednisone
  Arms: Thymectomy plus prednisone
Drug: prednisone alone — Prednisone regimen will be every other day, starting at 10mg. The dose will increase by 10mg every 2 days to a target dose.
  Other Names: prednisolone
  Arms: Prednisone alone

SUMMARY:
The purpose of this trial is to determine if thymectomy combined with prednisone therapy is more beneficial in treating non-thymomatous myasthenia gravis than prednisone therapy alone.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an autoimmune disease involving the thymus in which 85 percent of patients have antibodies to muscle acetylcholine receptors (AchR-Ab) that interfere with neuromuscular transmission. MG frequently causes severe disability that can be life-threatening. Thymectomy-a surgical procedure that removes thymus gland tissue from the chest cavity-has been an established therapy for non-thymomatous MG, or MG without thymoma, for more than 60 years (based on retrospective, non-randomized studies). Corticosteroids are now being used increasingly either as the sole treatment or in combination with thymectomy. Both therapies have associated adverse effects and indications for their use based on randomized trial data are lacking.

The purpose of this 5-year trial is to determine if the surgical procedure, extended transsternal thymectomy (ETTX), combined with prednisone therapy is more beneficial in treating individuals with non-thymomatous MG than prednisone therapy alone. More specifically, this study will determine 1) if ETTX combined with prednisone results in a greater improvement in myasthenic weakness, compared to prednisone alone; 2) if ETTX combined with prednisone results in a lower total dose of prednisone, thus decreasing the likelihood of concurrent and long-term toxic effects, compared to prednisone alone; and 3) if ETTX combined with prednisone enhances quality of life by reducing adverse events and symptoms associated with the therapies, compared to prednisone alone.

Learning that thymectomy results in a meaningful reduction of prednisone dosage or even full withdrawal or reduces side effects related to prednisone would support using the two treatments-thymectomy and prednisone-together. However, if no meaningful reduction of prednisone dosage or side effects is shown, the results would mean that using the two treatments together offers no advantages over prednisone treatment alone.

After an initial screening, study participants will be randomized either to undergo the surgical procedure ETTX and receive prednisone treatment, or to receive prednisone treatment alone without surgery. Participants will be followed for at least 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Male and female MG patients age greater than 18 and less than 65 years
* Onset of generalized MG within the last 5 years
* Positive serum anti-acetylcholine receptor binding antibodies (muscle acetylcholine receptors, AchRAb =/> 1.00 nmol/L. AchRAb levels of 0.50-0.99 nmol/L will be acceptable if there is another confirmatory test for MG, including single-fiber electromyography (EMG), repetitive nerve stimulation, or unequivocal edrophonium testing.)
* MGFA class II-IV at entry, using the MG Foundation of America (MGFA) classification, while receiving optimal anti-cholinesterase treatment with or without oral prednisone

Exclusion Criteria:

* Ocular MG without generalized weakness (MGFA Class I) or minimal weakness that would not require the use of corticosteroids
* Myasthenic weakness requiring intubation (MGFA Class IV) in the prior month
* Immunosuppressive therapy other than corticosteroids in the preceding year
* Medically unfit for thymectomy
* Chest CT evidence of thymoma.
* Pregnancy or lactation; contraindications to the use of corticosteroids, unless postmenopausal or surgically sterile. Women considering becoming pregnant during the period of the study are to be excluded.
* A serious concurrent medical, neurological or psychiatric condition that would interfere with thymectomy or subsequent clinical assessments
* Current alternate day dose of prednisone > than 1.5 mg/kg or 100 mg or the equivalent daily doses (> 0.75 mg/kg or 50 mg).
* Participation in another experimental clinical trial
* History of alcohol or drug abuse within the 2 years prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-06; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Cutter, PhD, Principal Investigator — University of Alabama at Birmingham School of Public Health, Department of Biostatistics; Gil Wolfe, MD, Principal Investigator — University of Buffalo, Jacobs School of Medicine and Biomedical Sciences; Henry Kaminski, MD, Principal Investigator — George Washington University School of Medicine and Health Sciences
Locations (70):
- United States (33):
  - University of Alabama at Birmingham, Department of Neurology, Sparks Center, Suite 350, 1720 7th Avenue South, Birmingham, Alabama
  - Data Coordination Center: University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Saint Joseph's Hospital and Medical Center, 350 W Thomas Rd, Phoenix, Arizona
  - University of Southern California, Doheny Institute, 1450 San Pablo St, Los Angeles, California
  - University of California Irvine, 101 The City Drive S, Bldg. 22 C, Route 13, Orange, California
  - California Pacific Medical Center, Castro St & Duboce Ave, San Francisco, California
  - University of Florida Jacksonville, Tower I, 8th Floor, 580 W. 8th ST., Jacksonville, Florida
  - University of Miami, 1120 NW 14th Street, Suite 1300, Miami, Florida
  - Emory University, 201 Dowman Dr, Atlanta, Georgia
  - Augusta University, 1120 15th St, Augusta, Georgia
  - Indiana University, Dept of Neurology, Regenstrief Health Center, 6th floor, 1050 Walnut St, Indiana University Medical Center, Indianapolis, Indiana
  - The University of Kansas Medical Center, 3901 Rainbow Blvd., Kansas City, Kansas
  - Brigham and Women's Hospital, 75 Francis Street, 5th Floor Tower, Boston, Massachusetts
  - Wayne State University School of Medicine, 4201 St Antoine, 8D UHC, Detroit, Michigan
  - William Beaumont Hospital, 3601 W. Thirteen Mile Road, Royal Oak, Royal Oak, Michigan
  - University of Minnesota, Department of Neurology, MMC 295, 420 Delaware St. S.E.,, Minneapolis, Minnesota
  - Mayo Clinic Rochester, 200 First St. SW, Rochester, Minnesota
  - St. Louis University, One North Grand St. Louis, St Louis, Missouri
  - Robert Wood Johnson University,, New Brunswick, New Jersey
  - Mount Sinai Hospital,1 Gustave L. Levy Pl, New York, New York
  - University of Rochester, 601 Elmwood Ave, Rochester, New York
  - Duke University, 200 Trent Dr, Durham, North Carolina
  - Case Western Reserve University, University Hospitals of Cleveland, 1100 Euclid Avenue, Cleveland, Ohio
  - The Ohio State University Wexmer Medical Center, Rm 461 Means Hall, The Ohio State University Medical Center,1654 Upham Dr., Columbus, Ohio
  - University of Texas Southwestern Medical Center, 5232 Harry Hines Blvd,, Dallas, Texas
  - University of Texas Medical Branch, 301 University Blvd, Galveston, Texas
  - Nerve and Muscle Center of Texas, 6624 Fannin St # 1670, Houston, Texas
  - University of Texas Health Science Center, Mail code 7883, 7703 Floyd Curl Drive, San Antonio, Texas
  - University of Vermont College of Medicine, Given Bldg C225, 89 Beaumont Avenue, Burlington, Vermont
  - University of Virginia, 1215 Lee St, Charlottesville, Virginia
  - University of Washington, 1410 NE Campus Pkwy, Seattle, Washington
  - West Virginia University, Dept of Neurology, WVU Eye Institute, Neurology Suite, 1 Stadium Drive,, Morgantown, West Virginia
  - Medical College of Wisconsin, 8701 Watertown Plank Road, Milwaukee, Wisconsin
- University of Buenis, Centro de Asistencia Docencia e Investigacion en Miastenia (CADIMI) Av. Forest 1146 - Ciudad Autonoma de Buenos Aires, Buenos Aires, Argentina
- Australia (2):
  - University of Sydney, Royal Prince Alfred Hospital and The University of Sydney, Sydney
  - University of Melbourne, Melbourne, The Royal Melbourne Hospital, Dept of Neurology, Royal Melbourne Hospital, Victoria
- Brazil (3):
  - Hospital de Base do Distrito Federal, Brasília
  - Universidade Federal do Parana, Curitiba
  - Federal University of Rio De Janeiro, Rio de Janeiro
- Canada (4):
  - University of Calgary, Heritage Medical Research Clinic Room 1132 3330 Hospital Dr NW, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Ottawa, The Ottawa Hospital General Campus, Division of Neurology, 501 Smyth Rd. Box 601, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec
- Hospital Del Salvador, Departamento de Ciencias Neurológicas, Universidad de Chile, Salvador 95 Of 416, Providencia, Santiago, Chile
- Germany (6):
  - University of Heidelberg, Seminarstraße 2, Mannheim, Baden-Wurttemberg
  - University of Regensburg, Dept. of Neurology, Universitätsstr. 84, D, Regensburg, Bavaria
  - University of Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Johannes-Gutenberg University, Klinikum der Johannes Gutenberg-Universität, Klinik und Poliklinik für Neurologie, Langenbeckstr, Mainz, Rhineland-Palatinate
  - University of Münster, Schlossplatz 2, Münster
  - University of Tübingen, Tübingen
- Italy (4):
  - National Neurological Institute "Carlo Besta", Myopathology and Immunology Unit, Dept of Neurology IV, Natl. Neurolog Inst. "C. Besta", Via Celoria, 11,, Milan
  - University of Rome "Sapienza", Rome
  - Catholic University, Universita Cattolica del Sacro Cuore, Largo Agostino Gemelli 8, e, Rome
  - University of Torino, Torino
- Japan (2):
  - Kanazawa University, Department of Neurology, Kanazawa University Hospital, 13-1 Takaramachi, Kanazawa, Ishikawa-ken
  - Nagasaki University, First Department of Internal Medicine,Graduate School of Biomedical Sciences,1-7-1,Sakamoto, Nagasaki, Kyushu
- Instituto Nacional de la Nutrición, México, Mexico
- Leiden University, Leiden, Netherlands
- Poland (2):
  - Medical University of Warsaw, Warsaw, Województwo
  - Institute of Tuberculosis and Lung Disease, Warsaw, Województwo
- Porto University, Serviço de Neurologia,Hospital Geral de Santo António, Largo Prof Abel Salazar, Porto, Portugal
- University of Cape Town, Division of Neurology E8-74, Groote Schuur Hospital,Observatory, Cape Town, South Africa
- H. Sant Pau, Universitat Autònoma de Barcelona, Neurology Department, Hospital Sta Creu i Sant Pau, C/Mas Casanovas no 90 4o pis 4o modul., Barcelona, Spain
- Fu-Jen Catholic University, No. 510, Zhongzheng Rd., Xinzhuang Dist, New Taipei City, Taiwan
- Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
- United Kingdom (5):
  - Queen Elizabeth University Hospital, Glasgow, Glasgow
  - Walton Centre for Neurology and Neurosurgery, Liverpool Heart and Chest Hospital, Liverpool. The Walton Centre for Neurology and Neurosurgery, Lower Lane, Fazakerley, Liverpool
  - University of Manchester, Oxford Road, Manchester
  - University of Oxford, Dept of Clinical Neurology, University of Oxford, Radcliffe Infirmary, Oxford
  - University of Sheffield, Western Bank, Sheffield

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Aban IB, Wolfe GI, Cutter GR, Kaminski HJ, Jaretzki A 3rd, Minisman G, Conwit R, Newsom-Davis J; Mgtx Advisory Committee. The MGTX experience: challenges in planning and executing an international, multicenter clinical trial. J Neuroimmunol. 2008 Sep 15;201-202:80-4. doi: 10.1016/j.jneuroim.2008.05.031. PMID 18675464
- [Result] Newsom-Davis J, Cutter G, Wolfe GI, Kaminski HJ, Jaretzki A 3rd, Minisman G, Aban I, Conwit R. Status of the thymectomy trial for nonthymomatous myasthenia gravis patients receiving prednisone. Ann N Y Acad Sci. 2008;1132:344-7. doi: 10.1196/annals.1405.014. PMID 18567886
- [Result] Minisman G, Bhanushali M, Conwit R, Wolfe GI, Aban I, Kaminski HJ, Cutter G. Implementing clinical trials on an international platform: challenges and perspectives. J Neurol Sci. 2012 Feb 15;313(1-2):1-6. doi: 10.1016/j.jns.2011.10.004. Epub 2011 Nov 1. PMID 22047648
- [Result] Kaminski HJ, Kusner LL, Wolfe GI, Aban I, Minisman G, Conwit R, Cutter G. Biomarker development for myasthenia gravis. Ann N Y Acad Sci. 2012 Dec;1275(1):101-6. doi: 10.1111/j.1749-6632.2012.06787.x. PMID 23278584
- [Result] Wolfe GI, Kaminski HJ, Aban IB, Minisman G, Kuo HC, Marx A, Strobel P, Mazia C, Oger J, Cea JG, Heckmann JM, Evoli A, Nix W, Ciafaloni E, Antonini G, Witoonpanich R, King JO, Beydoun SR, Chalk CH, Barboi AC, Amato AA, Shaibani AI, Katirji B, Lecky BR, Buckley C, Vincent A, Dias-Tosta E, Yoshikawa H, Waddington-Cruz M, Pulley MT, Rivner MH, Kostera-Pruszczyk A, Pascuzzi RM, Jackson CE, Garcia Ramos GS, Verschuuren JJ, Massey JM, Kissel JT, Werneck LC, Benatar M, Barohn RJ, Tandan R, Mozaffar T, Conwit R, Odenkirchen J, Sonett JR, Jaretzki A 3rd, Newsom-Davis J, Cutter GR; MGTX Study Group. Randomized Trial of Thymectomy in Myasthenia Gravis. N Engl J Med. 2016 Aug 11;375(6):511-22. doi: 10.1056/NEJMoa1602489. PMID 27509100
- [Derived] Lee I, Kuo HC, Aban IB, Cutter GR, McPherson T, Kaminski HJ, Sussman J, Strobel P, Oger J, Cea G, Heckmann JM, Evoli A, Nix W, Ciafaloni E, Antonini G, Witoonpanich R, King JO, Beydoun SR, Chalk CH, Barboi AC, Amato AA, Shaibani AI, Katirji B, Lecky BRF, Buckley C, Vincent A, Dias-Tosta E, Yoshikawa H, Waddington-Cruz M, Pulley MT, Rivner MH, Kostera-Pruszczyk A, Pascuzzi RM, Jackson CE, Verschuuren JJG, Massey JM, Kissel JT, Werneck LC, Benatar M, Barohn RJ, Tandan R, Mozaffar T, Conwit R, Minisman G, Sonett JR, Wolfe GI; MGTX study group. Minimal manifestation status and prednisone withdrawal in the MGTX trial. Neurology. 2020 Aug 11;95(6):e755-e766. doi: 10.1212/WNL.0000000000010031. Epub 2020 Jul 1. PMID 32611638
- [Derived] Wolfe GI, Kaminski HJ, Aban IB, Minisman G, Kuo HC, Marx A, Strobel P, Mazia C, Oger J, Cea JG, Heckmann JM, Evoli A, Nix W, Ciafaloni E, Antonini G, Witoonpanich R, King JO, Beydoun SR, Chalk CH, Barboi AC, Amato AA, Shaibani AI, Katirji B, Lecky BRF, Buckley C, Vincent A, Dias-Tosta E, Yoshikawa H, Waddington-Cruz M, Pulley MT, Rivner MH, Kostera-Pruszczyk A, Pascuzzi RM, Jackson CE, Verschuuren JJGM, Massey JM, Kissel JT, Werneck LC, Benatar M, Barohn RJ, Tandan R, Mozaffar T, Silvestri NJ, Conwit R, Sonett JR, Jaretzki A 3rd, Newsom-Davis J, Cutter GR; MGTX Study Group. Long-term effect of thymectomy plus prednisone versus prednisone alone in patients with non-thymomatous myasthenia gravis: 2-year extension of the MGTX randomised trial. Lancet Neurol. 2019 Mar;18(3):259-268. doi: 10.1016/S1474-4422(18)30392-2. Epub 2019 Jan 25. PMID 30692052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first enrollment of two patients started with July 26, 2006 and the last patient was recruited on November 28, 2012. Of the 126 randomized patients, 96 were from centers outside the US and 30 were from US centers.
Pre-assignment Details: After informed consent signed, 66 patients were randomized to extended transsternal thymectomy with prednisone treatment and 60 patients were assigned to take prednisone without surgery. Within the 126 subject that started, 15 dropped out before 3 year follow-up.
Groups:
- Thymectomy Plus Prednisone: Procedure: Extended Transsternal Thymectomy plus prednisone treatment
  thymectomy: The thymectomy had been performed as soon as possible after randomization.
- Prednisone Alone: Drug: prednisone alone protocol
  prednisone: Prednisone regimen had been taken every other day, starting at 10mg. The dose will increase by 10mg every 2 days to a target dose.
Period: Overall Study
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Started | 66 | 60
Completed | 60 | 51
Not Completed | 6 | 9
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Found to have invasive thymoma | 1 | 0
Not completed — Patient and family were not satisfied | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Thymectomy Plus Prednisone: Procedure: Extended Transsternal Thymectomy plus prednisone treatment
  thymectomy: The thymectomy will be performed as soon as possible after randomization.
- Prednisone Alone: Drug: prednisone alone protocol
  prednisone: Prednisone regimen will be every other day, starting at 10mg. The dose will increase by 10mg every 2 days to a target dose.
- Total: Total of all reporting groups
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone | Total
Number analyzed (Participants) | 66 | 60 | 126
Age, Continuous [Median (Full Range); unit: years] | 32 [18 to 63] | 33 [18 to 64] | 32 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 39 | 89
  Male | 16 | 21 | 37
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 4 | 10
  Black | 7 | 6 | 13
  Hispanic | 17 | 17 | 34
  Non-Hispanic | 31 | 30 | 61
  Other | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  Argentina | 10 | 11 | 21
  United States | 16 | 14 | 30
  Japan | 1 | 1 | 2
  United Kingdom | 2 | 2 | 4
  Thailand | 3 | 2 | 5
  Canada | 9 | 9 | 18
  Netherlands | 1 | 0 | 1
  Brazil | 3 | 2 | 5
  Poland | 1 | 1 | 2
  Italy | 6 | 4 | 10
  Mexico | 1 | 0 | 1
  South Africa | 4 | 4 | 8
  Australia | 2 | 2 | 4
  Chile | 5 | 5 | 10
  Germany | 2 | 3 | 5
Therapy at enrollment - Pyridostigimine [Number; unit: participants]
  Yes | 60 | 56 | 116
  No | 5 | 1 | 6
  Missing | 1 | 3 | 4
Therapy at enrollment - Glucocorticoid [Number; unit: participants]
  Yes | 49 | 47 | 96
  No | 16 | 10 | 26
  Missing | 1 | 3 | 4
Previous therapy - Intravenous immue globulin [Number; unit: participants]
  Yes | 12 | 13 | 25
  No | 53 | 44 | 97
  Missing | 1 | 3 | 4
Previous therapy - Plasma exchange [Number; unit: participants]
  Yes | 9 | 7 | 16
  No | 56 | 50 | 106
  Missing | 1 | 3 | 4
MGFA class [Number; unit: participants] — Class IIa. Predominantly affecting limb, axial muscles, or both. May also have lesser involvement of oropharyngeal muscles.
  Class IIb. Predominantly affecting oropharyngeal, respiratory muscles, or both. May also have lesser or equal involvement of limb, axial muscles, or both.
  Class III. Moderate weakness affecting muscles other than ocular muscles; may also have ocular muscle weakness of any severity.
  Class IV. Severe weakness affecting muscles other than ocular muscles; may also have ocular muscle weakness of any severity.
  Higher class was considered worse outcome.
  participants
    IIa | 25 | 25 | 50
    IIb | 18 | 14 | 32
    III | 21 | 20 | 41
    IV | 2 | 1 | 3
Duration of disease [Median (Full Range); unit: years] | 1.08 [0.02 to 4.41] | 1.14 [0.15 to 4.38] | 1.11 [0.02 to 4.41]
QMG score [Mean (Standard Deviation); unit: units on a scale] — Myasthenia Gravis (QMG) test. QMG total scores range from 0 to 39, with higher scores indicating more severe disease.
  units on a scale | 11.40 (5.12) | 12.35 (4.90) | 11.84 (5.02)
Prednisone use at baseline [Number; unit: participants]
  Yes | 49 | 47 | 96
  No | 16 | 10 | 26
  Missing | 1 | 3 | 4
Prednisone Dosage at baseline (mg) [Mean (Standard Deviation); unit: mg] — Prednisone dosage unit as mg, patient has been taken prednisone every other day
  mg | 43.43 (28.92) | 42.49 (23.52) | 42.97 (26.28)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average Quantitative Myasthenia Gravis Weakness Score Over 3 Years
Description: Myasthenia Gravis (QMG) test. QMG total scores range from 0 to 39 for a given visit, with higher scores indicating more severe disease. The time weighted average is a calculation that provides an integrated measure of the outcome over the time of followup. The denominator that was used to compute the time-weighted average for the Quantitative Myasthenia Gravis (QMG) score and the prednisone dose was the number of days from randomization to the last visit. Computations used the trapezoidal method where in the QMG score is multiplied by the number of days at this level from one visit to the next and added up over the entire followup experience and divided by the total number of days from randomization.
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Four participants in each group did not provide the information to enable calculation of the time-weighted Quantitative Myasthenia Gravis Weakness Score over 3 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 62 | 56
units on a scale | 6.15 (4.09) | 8.99 (4.93)

2. Primary Outcome: Time-weighted Average Alternate-day Prednisone Dose (mg) Measured Over 3 Years
Description: Participants reported alternate-day prednisone dose (mg) intake from baseline through withdrawn or completed 3 years follow up. The prednisone dosages had been weighted over the days of reporting period.
Time Frame: baseline, month 1 , 2 , 3, 4, 6 and every 3 months through 36 months
Population: Five participants in Thymectomy plus prednisone and 4 in Prednisone alone group did not provide the information to enable calculation of the time-weighted average alternate-day prednisone dose (mg) over 3 years.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 56
mg | 32 (23) | 54 (29)

3. Secondary Outcome: Subgroup Analyses of Time-weighted Average Quantitative Myasthenia Gravis Score by Prednisone Use at Enrollment
Description: Myasthenia Gravis (QMG) test. QMG total scores range from 0 to 39 for a given visit, with higher scores indicating more severe disease.
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Four participants in Thymectomy plus prednisone and 5 in Prednisone alone group did not provide information to enable the calculation of Time-weighted average Quantitative Myasthenia Gravis Score by prednisone use at enrollment over 3 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 62 | 55
units on a scale
  Not prednisone naïve: number analyzed (Participants) | 47 | 46
  Not prednisone naïve | 6.30 (3.89) | 9.10 (5.06)
  Prednisone naïve: number analyzed (Participants) | 15 | 9
  Prednisone naïve | 5.66 (4.79) | 8.84 (4.60)

4. Secondary Outcome: Subgroup Analyses of Time-weighted Average Quantitative Myasthenia Gravis Score by Sex
Description: as for outcome 3
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 62 | 56
units on a scale
  Female: number analyzed (Participants) | 46 | 38
  Female | 6.47 (4.13) | 9.73 (5.16)
  Male: number analyzed (Participants) | 16 | 18
  Male | 5.23 (3.95) | 7.45 (4.11)

5. Secondary Outcome: Subgroup Analyses of Time-weighted Average Quantitative Myasthenia Gravis Score by Age at Disease Onset
Description: as for outcome 3
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Four participants in each group did not provide the information to enable calculation of the time-weighted average Quantitative Myasthenia Gravis Weakness Score over 3 years. Another 2 participants in Thymectomy plus prednisone and 4 in Prednisone alone group did not provide the age at disease onset information.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 60 | 52
units on a scale
  Age (years) at Disease Onset < 40: number analyzed (Participants) | 42 | 34
  Age (years) at Disease Onset < 40 | 6.50 (4.41) | 9.60 (5.32)
  Age (years) at Disease Onset ≥ 40: number analyzed (Participants) | 18 | 18
  Age (years) at Disease Onset ≥ 40 | 5.33 (2.79) | 7.85 (3.50)

6. Secondary Outcome: Subgroup Analyses of Time-weighted Average Alternate-day Prednisone Dose (mg) by Prednisone Use at Enrollment
Description: as for outcome 2
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Five participants in Thymectomy plus prednisone and 4 in Prednisone alone group did not provide the information to enable calculation of time-weighted average alternate-day prednisone dose (mg) over 3 years. Another 1 in Prednisone alone group did not provide prednisone use at enrollment information.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 55
mg
  Not prednisone naïve: number analyzed (Participants) | 46 | 46
  Not prednisone naïve | 35 (25) | 56 (31)
  Prednisone naïve: number analyzed (Participants) | 15 | 9
  Prednisone naïve | 25 (17) | 45 (22)

7. Secondary Outcome: Subgroup Analyses of Time-weighted Average Alternate-day Prednisone Dose (mg) by Sex
Description: as for outcome 2
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 56
mg
  Female: number analyzed (Participants) | 45 | 37
  Female | 33 (25) | 54 (27)
  Male: number analyzed (Participants) | 16 | 19
  Male | 31 (18) | 55 (34)

8. Secondary Outcome: Subgroup Analyses of Time-weighted Average Average Alternate-day Prednisone Dose (mg) by Age at Disease Onset
Description: as for outcome 2
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Five participants in Thymectomy plus prednisone and 4 in Prednisone alone group did not provide the information to enable calculation of the time-weighted average alternate-day prednisone dose (mg) over 3 years. Another 2 in Thymectomy plus prednisone group and 4 in Prednisone alone group did not provide age at disease onset information.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 59 | 52
mg
  Age (Years) at Disease Onset < 40: number analyzed (Participants) | 41 | 33
  Age (Years) at Disease Onset < 40 | 35 (25) | 55 (30)
  Age (Years) at Disease Onset ≥ 40: number analyzed (Participants) | 18 | 19
  Age (Years) at Disease Onset ≥ 40 | 27 (18) | 49 (29)

9. Secondary Outcome: Number of Serious Adverse Events
Description: Number of participant who experienced at least one serious adverse events over 3 years: Thymectomy plus prednisone n=25 (out of 66); Prednisone alone n=33 (out of 60)
Time Frame: baseline to 3 years
Measure: Number; unit: events
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 25 | 33
events | 48 | 93

10. Secondary Outcome: Number of Patients With at Least One Serious Adverse Events
Description: as for outcome 9
Time Frame: baseline to 3 years
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
participants | 25 | 33

11. Secondary Outcome: Classification of Serious Adverse Events
Time Frame: baseline to 3 years
Population: One participant might had experienced more than one serious adverse event.
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 25 | 33
participants
  Life-threatening | 1 | 7
  Disability or incapacity | 8 | 2
  Medical or surgical intervention | 9 | 5
  Death | 0 | 1
  Complication due to thytmectomy | 1 | 0
  Hospitalization | 15 | 31

12. Secondary Outcome: Hospitalization for Exacerbation of Myasthenia Gravis
Time Frame: baseline to 2 years and baseline to 3 years
Population: Number of participants who had hospitalized over 2 and 3 years
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 15 | 31
participants
  Months 0-24 | 6 | 17
  Months 0-36 | 6 | 22

13. Secondary Outcome: Cumulative Number of Hospital Days
Description: Number who had hospitalization: Thymectomy plus prednisone n=15 (out of 66); Prednisone alone n=31 (out of 60)
Time Frame: baseline to 3 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 15 | 31
days | 8.4 (8.6) | 19.2 (24.5)

14. Secondary Outcome: Reason for Hospitalization According to Medical Dictionary for Regulatory Activities Term
Description: Number who had hospitalization: Thymectomy plus prednisone n=15 (out of 66); Prednisone alone n=31 (out of 60)
Time Frame: baseline to 3 years
Measure: Number; unit: events
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 15 | 31
events
  Gastrointestinal disorder | 2 | 2
  Hepatobiliary disorder | 0 | 1
  Infection or infestation | 4 | 7
  Injury, poisoning, or procedure complication | 2 | 0
  Metabolism or nutrition disorder | 1 | 0
  Nervous system disorder | 8 | 22
  Respiratory, thoracic, or mediastinal disorder | 1 | 2
  Surgical or medical procedure | 0 | 7
  Vascular disorder | 0 | 1

15. Secondary Outcome: Time-weighted Average Prescribed Alternate Day Prednisone Dose (mg)
Description: Physicians reported prescribed alternate-day prednisone dose (mg) intake from baseline through withdrawn or completed 3 years follow up. The prescribed prednisone dosages had been weighted over the days of reporting period.
Time Frame: baseline-day 20, month 1,2, 3, 4, 6 and every 3 months through 36 months
Population: Four participants in each group did not provide the information to enable calculation of the time-weighted average prescribed alternate-day prednisone dose (mg) over 3 years.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 62 | 56
mg | 34.3 (22.7) | 55.6 (29.4)

16. Secondary Outcome: Penalized Time-weighted Average Alternative Day Prednisone Dose (mg; Method 1: Penalized Using Maximum Dose Before Azathioprine)
Description: For each participant who took azathioprine, we penalized them by taking the maximum dose of prednisone before azathioprine was added. We then applied the same method to compute the time-weighted alternative day prednisone dose from baseline, month 3, 4, 6 and every 3 months through 36 months.
Time Frame: baseline, month 3, 4, 6 and every 3 months through 36 months
Population: Five participants in Thymectomy plus prednisone and 4 in Prednisone alone group did not provide the information to enable calculation of the penalized time-weighted average alternate-day prednisone dose (mg) over 3 years.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 56
mg | 34.4 (28.2) | 64.4 (40.8)

17. Secondary Outcome: Penalized Time-weighted Average Alternative Day Prednisone Dose (mg; Method 2: Penalized Using Dose at Time of Starting Azathioprine)
Description: For each participant who took azathioprine, we penalized them by taking the prednisone dose at the time azathioprine commenced. We then applied the same method to compute the time-weighted alternative day prednisone dose from baseline, month 3, 4, 6 and every 3 months through 36 months.
Time Frame: baseline, month 1 , 2 , 3, 4, 6 and every 3 months through 36 months
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 56
mg | 33.3 (27.2) | 57.9 (36.9)

18. Secondary Outcome: Time-Weighted Average MG Activity of Daily Living (MG-ADL)
Description: MG Activity of Daily Living total scores range from 0 to 24, with the lower scores indicating better daily living quality of life.
Time Frame: baseline, month 4, 6 and every 3 months through 36 months
Population: Five participants in each group did not provide the information to enable calculation of the time-weighted average MG activity of daily life over 3 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 61 | 55
units on a scale | 2.24 (2.09) | 3.41 (2.58)

19. Secondary Outcome: Time-Weighted Average MG Activity of Daily Living (MG-ADL) at Month 12, 24, and 36
Description: MG Activity of Daily Living total scores range from 0 to 24 by visit, with the lower scores indicating better daily living quality of life.
Time Frame: Month 12, 24, and 36
Population: Participants were in and out at month 12, 24 and 36 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
units on a scale
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 1.92 (2.73) | 3.33 (3.40)
  Month 24: number analyzed (Participants) | 59 | 53
  Month 24 | 2.02 (2.78) | 3.11 (2.93)
  Month 36: number analyzed (Participants) | 59 | 51
  Month 36 | 2.14 (2.92) | 2.69 (2.80)

20. Secondary Outcome: Azathioprine Use
Time Frame: baseline to 3 years
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 65 | 58
participants | 11 | 28

21. Secondary Outcome: Plasma Exchange Use
Time Frame: baseline to 3 years
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 65 | 58
participants | 10 | 9

22. Secondary Outcome: Intravenous Immunoglobulin Use
Time Frame: baseline to 3 years
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 65 | 58
participants | 11 | 23

23. Secondary Outcome: Minimal Manifestation (MM) Status at Month 12, 24 and 36
Description: Number of participants who were in minimal manifestation status at month 12, 24 and 36.
Time Frame: Month 12, 24 and 36
Population: Number analyzed: Thymectomy plus prednisone: n=61 (Month 12), 59 (Month 24) , and 58 (Month 36); Prednisone alone n=54 (Month 12), 53 (Month 24), and 51 (Month 36)
Measure: Number; unit: participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
participants
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 41 | 20
  Month 24: number analyzed (Participants) | 59 | 53
  Month 24 | 39 | 20
  Month 36: number analyzed (Participants) | 58 | 51
  Month 36 | 39 | 24

24. Secondary Outcome: Cumulative Days in Hospital for Myasthenia Gravis Exacerbation
Description: Number of patients with MG exacerbation: Thymectomy plus prednisone=6 (out of 66); Prednisone alone=17 (out of 60)
Time Frame: baseline to 2 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 6 | 17
days | 5.5 (2.9) | 26.4 (28.9)

25. Secondary Outcome: Cumulative Days in Hospital for Myasthenia Gravis Exacerbation
Description: Number of patients with MG exacerbation: Thymectomy plus prednisone=6 (out of 66); Prednisone alone=22 (out of 60)
Time Frame: baseline to 3 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 6 | 22
days | 8.7 (7.7) | 22.5 (27.1)

26. Secondary Outcome: Short Form-36 Standardized Physical Component
Description: Range from 0 to 100, the higher the physical component value, the better the mental health.
Time Frame: Month 0, Month 12, Month 24 and Month 36
Population: Participants were in and out by visit.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
units on a scale
  Month 0: number analyzed (Participants) | 65 | 58
  Month 0 | 41.4 [18.2 to 60.0] | 37.9 [13.5 to 64.3]
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 48.4 [11.5 to 64.4] | 44.4 [21.2 to 58.8]
  Month 24: number analyzed (Participants) | 59 | 53
  Month 24 | 50.3 [11.2 to 60.5] | 43.0 [25.3 to 59.6]
  Month 36: number analyzed (Participants) | 58 | 50
  Month 36 | 48.2 [9.8 to 61.8] | 44.2 [20.4 to 58.9]

27. Secondary Outcome: Short Form-36 Standardized Mental Component
Description: Range from 0 to 100, the higher the mental component value, the better the mental health.
Time Frame: Month 0, Month 12, Month 24 and Month 36
Population: Participants were in and out by visit.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
units on a scale
  Month 0: number analyzed (Participants) | 65 | 58
  Month 0 | 49.1 [14.6 to 65.3] | 46.2 [22.4 to 70.7]
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 39.1 [17.6 to 66.7] | 41.7 [7.6 to 64.4]
  Month 24: number analyzed (Participants) | 59 | 53
  Month 24 | 49.9 [14.4 to 62.3] | 46.7 [21.3 to 69.1]
  Month 36: number analyzed (Participants) | 58 | 50
  Month 36 | 51.7 [29.9 to 65.1] | 48.2 [24.1 to 69.2]

28. Secondary Outcome: Treatment Associated Complications (TAC)
Description: Treatment associated complications measured complications occurred by myasthenia gravis patients. Report number of participant with at least one complications by each visit.
Time Frame: Month 0, 1, 2, 3, 4 then every 3 months through Month 36
Population: Participants were in and out by each visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
Participants
  Month 0: number analyzed (Participants) | 65 | 58
  Month 0 | 22 | 17
  Month 1: number analyzed (Participants) | 58 | 56
  Month 1 | 15 | 15
  Month 2: number analyzed (Participants) | 61 | 55
  Month 2 | 22 | 20
  Month 3: number analyzed (Participants) | 61 | 55
  Month 3 | 21 | 16
  Month 4: number analyzed (Participants) | 62 | 56
  Month 4 | 23 | 23
  Month 6: number analyzed (Participants) | 61 | 55
  Month 6 | 21 | 22
  Month 9: number analyzed (Participants) | 61 | 54
  Month 9 | 37 | 26
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 35 | 28
  Month 15: number analyzed (Participants) | 60 | 53
  Month 15 | 29 | 24
  Month 18: number analyzed (Participants) | 59 | 53
  Month 18 | 28 | 24
  Month 21: number analyzed (Participants) | 60 | 52
  Month 21 | 22 | 20
  Mpnth 24: number analyzed (Participants) | 59 | 53
  Mpnth 24 | 28 | 23
  Mpnth 27: number analyzed (Participants) | 61 | 53
  Mpnth 27 | 25 | 17
  Month 30: number analyzed (Participants) | 58 | 53
  Month 30 | 23 | 19
  Month 33: number analyzed (Participants) | 61 | 52
  Month 33 | 24 | 23
  Month 36: number analyzed (Participants) | 59 | 51
  Month 36 | 23 | 23

29. Secondary Outcome: Treatment Associated Symptoms (TAS)
Description: Treatment associated symptoms measured myasthenia gravis symptoms such as back pain and/or bruises. Report number of participant with at least one treatment associated symptoms by each visit.
Time Frame: Month 0, 1, 2, 3, 4 then every 3 months through Month 36
Population: Patients were in and out by visit
Measure: Count of Participants; unit: Participants
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Number analyzed (Participants) | 66 | 60
Participants
  Month 0: number analyzed (Participants) | 65 | 57
  Month 0 | 63 | 53
  Month 1: number analyzed (Participants) | 58 | 56
  Month 1 | 55 | 52
  Month 2: number analyzed (Participants) | 61 | 55
  Month 2 | 61 | 53
  Month 3: number analyzed (Participants) | 61 | 55
  Month 3 | 60 | 54
  Month 4: number analyzed (Participants) | 62 | 56
  Month 4 | 59 | 54
  Month 6: number analyzed (Participants) | 61 | 55
  Month 6 | 60 | 53
  Month 9: number analyzed (Participants) | 61 | 54
  Month 9 | 59 | 50
  Month 12: number analyzed (Participants) | 61 | 54
  Month 12 | 56 | 52
  Month 15: number analyzed (Participants) | 60 | 53
  Month 15 | 56 | 51
  Month 18: number analyzed (Participants) | 59 | 53
  Month 18 | 52 | 51
  Month 21: number analyzed (Participants) | 60 | 52
  Month 21 | 52 | 50
  Mpnth 24: number analyzed (Participants) | 59 | 53
  Mpnth 24 | 52 | 51
  Mpnth 27: number analyzed (Participants) | 61 | 53
  Mpnth 27 | 50 | 50
  Month 30: number analyzed (Participants) | 58 | 53
  Month 30 | 49 | 50
  Month 33: number analyzed (Participants) | 61 | 51
  Month 33 | 51 | 48
  Month 36: number analyzed (Participants) | 60 | 51
  Month 36 | 49 | 47

ADVERSE EVENTS:
Time Frame: Adverse events were reported from baseline to 3 years
Description: There were two groups: 60 patients who received prednisone only and 66 patients had thymectomy plus prednisone
Arm/Group | Thymectomy Plus Prednisone | Prednisone Alone
Serious Adverse Events (participants affected / at risk) | 25/66 | 33/60
Other Adverse Events (participants affected / at risk) | 55/66 | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymectomy Plus Prednisone (N=66) | Prednisone Alone (N=60)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 3 (4)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Incision site cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (2) | 3 (3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 6 (7) | 22 (43)
Myasthenia gravis crisis (Nervous system disorders) | 4 (6) | 10 (13)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Diaphragm muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eye operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Supportive care (Surgical and medical procedures) | 0 (0) | 1 (1)
Thoracotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Thymectomy (Surgical and medical procedures) | 0 (0) | 7 (7)
Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thymectomy Plus Prednisone (N=66) | Prednisone Alone (N=60)
Cataract (Eye disorders) | 4 (14) | 7 (20)
Glaucoma (Eye disorders) | 5 (22) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (6) | 4 (8)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Liver function test abnormal (Investigations) | 2 (2) | 3 (3)
Abnormal weight gain (Metabolism and nutrition disorders) | 32 (184) | 31 (141)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (41) | 9 (44)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 15 (43) | 4 (9)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Mental disorder (Psychiatric disorders) | 4 (4) | 5 (8)
Sleep disorder (Psychiatric disorders) | 25 (86) | 22 (67)
Rash (Skin and subcutaneous tissue disorders) | 21 (58) | 24 (48)
Scab (Skin and subcutaneous tissue disorders) | 11 (44) | 2 (2)
Hypertension (Vascular disorders) | 16 (53) | 16 (55)

LIMITATIONS AND CAVEATS:
Potential weakness of this trial include the single-blinded and pill count methodology.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days